CLINICAL TRIAL: NCT02789605
Title: Treatment of Idiopathic and Recurrent Aphthous Stomatitis by a Probiotic, the Lactobacillus Rhamnosus Lcr35® : a Randomized, Double Blind and Placebo-controlled Trial
Brief Title: Effectiveness and Safety of Lactobacillus Rhamnosus Lcr35® in the Treatment of Recurrent Aphthous Stomatitis
Acronym: Aphtose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-PP-13
Record Dates: First submitted 2016-04-14; First posted 2016-06-03 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2019-12

CONDITIONS: Aphthous Stomatitis
Keywords: Aphthous Stomatitis [C07.465.864.750]
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacilor (Experimental): Patient receiving Lactobacillus rhamnosus Lcr35®, orally taken, 4 times a day, during 3 months
  Interventions: Drug: Bacilor
- Placebo (Placebo Comparator): Patient receiving placebo, orally taken, 4 times a day, during 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bacilor — Patient receiving Lactobacillus rhamnosus Lcr35®, orally taken, 4 times a day, during 3 months. Then all patients will be then followed up for 3 additional months without treatment.
  Arms: Bacilor
Drug: Placebo — Patients of group B will took the placebo similarly at the Lactobacillus rhamnosus Lcr35® orally . All patients will be then followed up for 3 additional months without treatment.
  Arms: Placebo

SUMMARY:
Recurrent aphthous stomatitis (RAS) is a frequent condition characterized by recurrent and painful oral ulcers with unknown pathophysiology. Recent studies suggest that a dysregulation of the oral microbiota may be implicated. Currently, therapies for RAS are limited by severe side effects or inconstant effectiveness. The aim of this study is to assess the effectiveness and safety of a probiotic, the Lactobacillus rhamnosus Lcr35® , in the treatment of RAS. A placebo-controlled, parallel study will be conducted in 40 subjects with RAS. Treatment consisted on the administration of the daily probiotics or placebo during 3 months.All patients will be then followed up for additional 3months without treatment. The main outcome measure will be the number of occurring aphtae.

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is the most common chronic disease of the oral cavity, affecting 5-25% of the population. This condition is characterized by recurrent and painful oral ulcers. The discomfort of RAS can impact negatively on quality of life that is why the therapeutic demand is strong. Currently, there is no curative treatment for RAS, and suspensive treatments such as colchicine and thalidomide are no definitive or can induce severe side effects. The pathophysiology of RAS remains largely unknown. Recent studies suggest that a dysregulation of the oral microbiota may be implicated. Increasing data underline the potential interest of using probiotics in conditions due to microbiota disorder. To the best of our knowledge, no study has evaluated the effectiveness of probiotic in RAS. The main objective of this double blind clinical trial is to evaluate the effectiveness and safety of a probiotic, the Lactobacillus rhamnosus Lcr35®, in the treatment of RAS in adults. 40 patients suffering from minor RAS for 6 months will be included and randomly assigned to 2 group of 20. Patients of group A will took the Lactobacillus rhamnosus Lcr35® orally daily for 3 months and patients of group B will took the placebo similarly. All patients will be then followed up for 3 additional months without treatment. The primary outcome measure will be the monthly number of aphthae occurring during the 3 months of treatment. The secondary outcomes measures will be the monthly number of aphthae occurring during the 3 months of follow up, the pain reduction, the impact on quality of life according to the OHIP-14 score and the side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 year-old or more
* Recurrent idiopathic aphtous stomatitis with at least one new lesion per month during the past 6 months.

Exclusion Criteria:

* Symptomatic aphtosis associated with Crohn or Behcet disease
* Concomitant use of probiotic for any other reason
* Systemic use of colchicine or steroids or immunosuppressive drugs during the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
number of aphtae | from baseline at 3 months
  The number of aphtae

SECONDARY OUTCOMES:
Quality of life | At 3 months
  the impact on quality of life according to the OHIP-14 score
Satisfaction patient | At 3 months
  the satisfaction of the patients about effectiveness and safety of the treatments by EVA.

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — CHU de Nice, Hôpital Archet, Dermatologie
Locations (1):
- CHU de NIce - Dermatologie, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No